CLINICAL TRIAL: NCT06481293
Title: Tackling Dry Socket Via Dual Wavelength Laser Diode Therapy in Smokers: A Randomized Controlled Trial.
Brief Title: Tackling Dry Socket Via Laser Therapy in Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Badr University (Other)
Responsible Party: Principal Investigator, Reham Alaa, lecturer of physical therapy, Badr University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BUC-IACUC-231015-42
Record Dates: First submitted 2024-06-25; First posted 2024-07-01 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Alveolar Osteitis
Keywords: Diode laser; Dry socket
MeSH Terms: conditions — Dry Socket

STUDY DESIGN:
Intervention Model Description: The study included two groups. One group receives dual wavelength laser diode therapy and the other group receives topical aveogyl dressing.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 received diode laser therapy
  Interventions: Device: Diode laser therapy
- group 2 (Experimental): Group 2 received topical application of aveogl dressing
  Interventions: Combination Product: Alveogyl dressing

INTERVENTIONS:
Device: Diode laser therapy — Dual wavelength laser diode therapy device
  Arms: Group 1
Combination Product: Alveogyl dressing — Alveogyl is a haemostatic-analgesic alveolar dressing
  Arms: group 2

SUMMARY:
This study examines the efficiency of diode laser therapy to manage dry sockets after tooth extraction.

DETAILED DESCRIPTION:
The study compares the efficiency of diode laser therapy and using only alveogyl to accelerate the healing of dry sockets after tooth extraction in smokers. Smoker patients with dry sockets were enrolled randomly into two different groups. Group 1 received dual wavelength laser diode therapy, three times per week. While group 2 received only a topical application of alveogl. The treatment lasted for two consecutive weeks. The treatment efficiency was evaluated by measuring the volume of the socket using the syringe method. The pain level was measured by the visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Smokers patient

Exclusion Criteria:

* Females on contraceptives.
* Diabetic patients
* Hepatitis C virus patients
* Patients on corticosteroids
* Patients with renal diseases
* Anemic patients

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Socket volume | 2 weeks
  measured through the volumetric measurement method using a syringe filled with saline

SECONDARY OUTCOMES:
Pain level | 2 weeks
  measured by the visual analogue scale(VAS). It include score from 0 to 10 in which 10 indicates the worst pain level and 0 indicates no pain

CONTACTS AND LOCATIONS:
Overall Officials: reham Elkalla, lecturer, Principal Investigator — Badr University in Cairo
Locations (1):
- Badr University in Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No